CLINICAL TRIAL: NCT06994156
Title: Diagnostic and Prognostic Salivary Biomarkers in Chronic Muscle Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Eastmaninstitutet (Other)
Responsible Party: Principal Investigator, Hajer Jasim, Principal Investigator, Karolinska Institutet
Other Study IDs: DNR 2023-03570-01
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: TMD/Orofacial Pain; Fibromyalgia (FM)
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Muscle pain: Patients diagnosed with myogenious TMD and patients diagnosed with Fibromyalgia according to ACR 1990/2016
- Control: Matched healthy controls

SUMMARY:
A large proportion of the adult population worldwide currently lives with chronic muscle pain, with more than half of those affected experiencing pain localized to the face and jaw. This means that approximately 10-15% of the adult population is affected. Living with chronic muscle pain impacts many aspects of life, significantly affecting both the individual's quality of life and well-being as well as that of their close relations.

As with other chronic pain conditions, researchers agree that multiple factors contribute to the development and aggravation of the condition. The aim of this project is to identify proteins in saliva that are involved in the disease process of chronic muscle pain, in order to better understand the underlying mechanisms, improve prognosis assessment, and ultimately develop more effective treatments.

The project includes patients with localized chronic jaw muscle pain, those with generalized chronic pain (fibromyalgia), and pain-free individuals in a matched control group. Validated questionnaires are used to assess pain, including measures of physical and emotional function, followed by a clinical examination. Chewing-stimulated saliva is selected for sampling based on previous studies from the research group, and blood samples are collected from all participants. Proteins involved in metabolism, stress, and immunity will be analyzed, building on prior research conducted by the group. Patients will undergo conventional orofacial pain treatment and will later be followed up with new samples to study changes in protein expression following successful treatment.

Chronic muscle pain is one of the leading causes of work incapacity and long-term sick leave. This project combines clinical examinations with advanced biomedical analysis methods to investigate the role of specific proteins in disease development. The goal is to identify proteins involved in pain mechanisms to improve diagnostics and enable personalized treatments. In the short term, this could lead to faster and more accurate diagnoses and the development of new treatment strategies, which would reduce pain intensity and work incapacity, ultimately benefiting both individuals and society.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of myalgia or myofascial pain with referral according to the DC/TMD Axis I
* Diagnosis of fibromyalgia according to ACR 1990 or ACR 2016 criteria
* Minimum pain intensity of 30 on a 100 mm visual analogue scale (VAS)

Exclusion Criteria

* Diagnosed systemic muscular or joint diseases (except for fibromyalgia)
* Whiplash-associated disorder
* Migraine
* Neurological disorders
* Neuropsychiatric disorders
* Diseases of the salivary glands (e.g., sialadenitis, salivary gland tumours)
* Pregnancy and lactation
* Obesity
* Use of analgesics within the last 24 hours
* Oral complaints such as oral dryness
* Mucosal lesions in the oral cavity
* Fewer than 22 natural teeth
* Extensive prosthodontic rehabilitations
* Poor oral hygiene
* Hyposalivation
* Oral diseases (periodontal diseases and mucosal pain or ulcerations)
* Extensive dental abrasion

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Participants will be recruited through advertisement and from patients referred to the specialist clinic for orofacial pain and jaw function at the University Dental Clinic at Karolinska Institute (Huddinge, Sweden) and at Eastman Institutet, Folktandvården Stockholm.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in salivary protein expression levels | 7 months
  Change in salivary protein expression levels (e.g., inflammation-, stress-, or metabolism-related biomarkers) before and after conventional orofacial pain treatment,

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Department of Dental Medicine, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Undecided